CLINICAL TRIAL: NCT05095025
Title: PENG Block for Patients Undergoing Neck of Femur (NOF) Fracture Surgery: a Dose Finding Study
Brief Title: PENG: an Estimation of ED50 in Neck of Femur Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Brian Declan O'Donnell, Consultant Anaesthesiologist, University College Cork
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PENG Dose 1
Record Dates: First submitted 2021-09-20; First posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Hip Fractures; Pain, Acute
Keywords: bupivacaine; dose; PENG Block; Regional Anesthesia
MeSH Terms: conditions — Hip Fractures; Acute Pain | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Using a sequential step-up, step-down dosing model the dose of bupivacaine administered will be determined by the response of the preceding patient. Each participant will receive a total injectate volume of 20ml. Based upon the published efficacy literature, the starting dose of bupivacaine will be 50mg. The dose of bupivacaine will be adjusted by 5mg up or down based on the outcome (analgesic success or failure) of each subsequent participant.
Masking Description: The assessor and the patient will be unaware of the dose of bupivacaine administered. The bupivacaine solution will be prepared by an investigator other than those involved in the performance of the PENG block or the assessment of block outcome.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bupivacaine dose finding (Experimental): Sequential up and down dose modification based on the outcome of the intervention in the preceding participant
  Interventions: Drug: Bupivacaine Hydrochloride 20ml injectate

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride 20ml injectate — Sequential dosing, starting at 50mg with 5mg increments based on the outcome of the preceding participant
  Other Names: Sequential up and down dosing

SUMMARY:
The effective dose of local anaesthetic used in PENG blocks to achieve analgesia in patients with fractured neck of femur is unknown. It is planned to address this question using a dixon/massey sequential dosing methodology to establish the ED50 of 0.25% Bupivacaine.

DETAILED DESCRIPTION:
Neck of femur (NOF) fracture is a common presentation to the emergency department, particularly in the older population. 77,210 NOF fractures were recorded in the UK and Ireland in 2018 and the number of cases is projected to increase as life expectancy improves. NOF fracture is associated with a high social and economic cost, estimated to cost €45 million annually in Ireland with significant effects on patients' quality of life

The latest Irish Hip Fracture Database (IHFD) report from 2019 detailed 3,701 NOF fractures in patients over 60 years of age in Ireland. These patients occupied 72,314 acute hospital bed days nationally and 437 of these patients attended CUH. This frail and vulnerable group had an average age of 81 and many people suffered numerous co-morbid conditions. This population of patients is therefore at significant risk of complications and require multidisciplinary input to optimise clinical outcome

From a patient's perspective, NOF fracture is a very painful condition, requiring early surgical fixation. It is associated with significant morbidity and mortality. The 30-day mortality for this condition has improved recently. This has likely multifactorial, in part due to the introduction of clinical guidelines, national audits, a focus on processes and changes in how hip fracture care is funded. However, 5% of patients who sustained a hip fracture in Ireland in 2019 died. An additional 4% of patients required new admission to a nursing home following this fracture and a further 13% required convalescent care.

These patients are also particularly at risk for under treatment of pain. Contraindications to many commonly used analgesics such as non-steroidal anti-inflammatory drugs (NSAIDs) exist in this population, including renal dysfunction in 40%. Older adults suffer more adverse effects from opiate analgesia such as nausea, vomiting, constipation, drowsiness and respiratory complications. This population also have a 25% incidence of cognitive impairment which may make communication and assessment of their pain more challenging.

Regional anaesthesia (RA) has been extensively researched in this group of patients with a view to improving the quality of pain relief while reducing the side effects of analgesic medications used. In 2017, a Cochrane review on RA in the management of patients with NOF fractures concluded that there was high quality evidence that RA reduces pain on movement within 30 minutes after block placement and reduces opioid consumption and moderate quality evidence that RA reduces the incidence of pneumonia, time to first mobilization and cost.

Widespread use of RA on admission to hospital and in the early postoperative period is also supported by the latest Association of Anaesthetists' (AoA)guideline: "Guideline for the management of hip fractures 2020". In this, femoral or fascia iliaca blocks are recommended as pericapsular nerve group (PENG) blocks have not yet been compared with these more established blocks in trials. It is also recommend that general anaesthesia or spinal anaesthesia should be routinely supplemented with RA and state that there is little evidence at present for continuous catheter techniques which may delay remobilisation.

Single injection RA blocks are limited by their short duration which can be prolonged by continuous catheter techniques. A study from Cork University Hospital published in 2012 demonstrated more effective perioperative analgesia, reduced opiate consumption and improved patient satisfaction when continuous femoral nerve blockade was compared with a standard opiate based regime in patients with NOF fractures for up to 54 hours on passive movement and up to 42 hours at rest. However, femoral nerve blockade can be associated with weakness of the quadriceps muscle, possibly reducing early postoperative mobility and increasing the risk of falls. A study of healthy volunteers demonstrated a significant reduction in quadriceps strength and balance scores following femoral nerve blockade. Another study suggested a causal relationship between continuous peripheral nerve blocks and falls after hip and knee arthroplasty.

The pericapsular nerve group (PENG) block, first described in 2018, is a RA technique which aims to provide analgesia for patients with NOF fractures by blocking sensory branches of the femoral nerve, obturator nerve and accessory obturator nerve to the anterior hip capsule. This may improve analgesia to the NOF fracture site compared with femoral nerve blockade, while sparing the branches of the femoral nerve which supply motor innervation to the quadriceps muscle, thereby lessening muscle weakness. A published dissection of an embalmed cadaver injected with 10ml and 20ml of dye via PENG block demonstrated that both volumes spread to the articular branches of the femoral, obturator and accessory obturator nerves but there is no published data in patients.

Continuous catheter techniques have also been described for this block.

This study aims to measure the dose of bupivacaine required to provide adequate analgesia at 30 minutes. As described above, there is a lack of available data on the effective dose. Given the proposed mechanism and the demonstrated spread of local anaesthetic injected via PENG block, as well as published results from case series, it is plausible that PENG blocks produce superior analgesia to the currently used femoral blocks and fascia iliaca blocks. For similar reasons, PENG blocks are likely associated with significantly less leg weakness compared with femoral nerve blocks; there are 2 reported cases in the published literature, both attributed to inadvertent femoral block. Finally, the latest AoA guidelines cite a lack of evidence and delayed remobilization as reasons against using continuous catheter techniques. Lack of motor weakness is a proposed benefit of this block and the possibility of improved pain relief postoperatively is likely to enhance a patient's remobilisation, increasing the importance of this study.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for operative repair of hip fracture
* Patient age 18 years or more
* ASA I - III

Exclusion Criteria:

* Patient refusal
* Coagulopathy
* Local infection
* Allergy to Local Anaesthetics
* Significant cognitive impairment (4AT score>=4 or otherwise unable to provide consent)
* Previous RA procedure within 24hours with ongoing analgesia
* Weight <50kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Analgesic success | 30 minutes
  Verbal rated pain score of ≤3/10 30 minutes after the administration of a predetermined dose of bupivacaine via a continuous PENG catheter

SECONDARY OUTCOMES:
Analgesic failure | 30 minutes
  Verbal rated pain score of ≥ 3/10 30 minutes after the administration of a predetermined dose of bupivacaine via a continuous PENG catheter

OTHER OUTCOMES:
Effective dose in 50 % of participants | 30 minutes
  The dose of bupivacaine which results in 5 independent pairs of participants with sequential analgesic block success and failure.

CONTACTS AND LOCATIONS:
Overall Officials: Brian O'Donnell, MD, Principal Investigator — UCC
Locations (1):
- Cork University Hospital, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No